CLINICAL TRIAL: NCT00889850
Title: Open, Randomised, Single-Dose, 2x2-Way Cross-Over Comparative Oral Bioavailability Study in Healthy Adult Male Subjects Under Fasted Conditions (Block I) and Under Fed Conditions (Block II); Comparison of 40 mg Esomeprazole Mepha Capsules (Test) With 40 mg Esomeprazole INexium MUPS Tablets (Reference)
Brief Title: Esomeprazole Bioavailability Study With 40 mg Oral Single Dose Fasted and Fed Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mepha Ltd. (Industry)
Collaborators: SocraTec R&D GmbH (Other); SocraMetrics GmbH (Industry)
Responsible Party: Sabine Galliker, Mepha
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: ESO 001.2009; SocraTec: 1216es09ct; EudraCT: 2009-010941-29
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Healthy; Bioavailability; Bioequivalence; Esomeprazole; Bioavailability, Therapeutical Indication Not Studied
MeSH Terms: interventions — major urinary proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Oral fasted administration of one capsule of 40 mg Esomeprazole Mepha (Mepha Ltd., Switzerland)
  Interventions: Drug: 40 mg Esomeprazole Mepha (Mepha Ltd., Switzerland)
- 2 (Active Comparator): Oral fasted administration of one tablet of INexium 40 mg MUPS tablets (AstraZeneca, France)
  Interventions: Drug: INexium 40 mg MUPS tablets (AstraZeneca, France)
- 3 (Active Comparator): Oral fed administration of one capsule of 40 mg Esomeprazole Mepha (Mepha Ltd., Switzerland)
  Interventions: Drug: 40 mg Esomeprazole Mepha (Mepha Ltd., Switzerland)
- 4 (Active Comparator): Oral fed administration of one tablet of INexium 40 mg MUPS tablets (AstraZeneca, France)
  Interventions: Drug: INexium 40 mg MUPS tablets (AstraZeneca, France)

INTERVENTIONS:
Drug: 40 mg Esomeprazole Mepha (Mepha Ltd., Switzerland) — 40 mg esomeprazole, single dose administration under fasted and fed condition
  Other Names: Test
  Arms: 1; 3
Drug: INexium 40 mg MUPS tablets (AstraZeneca, France) — 40 mg esomeprazole, oral single dose administration under fasted and fed condition
  Other Names: Reference
  Arms: 2; 4

SUMMARY:
The present study will be conducted in order to compare the bioavailability of 40 mg Esomeprazole Mepha (Mepha Ltd., Switzerland) and of INexium 40 mg MUPS tablets (AstraZeneca, France) under single dose fasted and fed conditions.

The study will be conducted as a combined single dose study under fasted and fed conditions in a 2x2-period cross-over design with a wash out phase of at least 6 treatment-free days between administrations.

DETAILED DESCRIPTION:
* The primary objective of the single dose fasted part of the study is to compare the rate and extent of absorption of esomeprazole from 40 mg Esomeprazole Mepha capsules (Test) with 40 mg Esomeprazole INexium MUPS tablets (Reference) after single dose administration under fasted conditions, determined by use of AUC0-tlast and Cmax obtained from esomeprazole plasma concentrations.
* The primary objective of the single dose fed in combination with the fasted part of the study is to compare the maximum concentration of esomeprazole determined after 40 mg Esomeprazole Mepha capsules (Test) single dose administration under fed conditions in comparison with 40 mg Esomeprazole INexium MUPS tablets (Reference) after single dose administration under fasted and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subject has to:

  1. be Caucasian male
  2. be aged between 18-55 years, inclusive
  3. have a body-mass index (BMI): ≥ 19 kg/m² and ≤ 27 kg/m²
  4. be considered to be healthy on the basis of extensive pre-study eligibility assessment
  5. be a non-smoker or an ex-smoker for at least 1 month
  6. be willing and capable to confirm written consent to enrolment after ample information has been provided

Exclusion Criteria:

* Subjects cannot be included if they match any of the following exclusion criteria:

  1. existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the drug, i.e. impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhoea or conditions associated with total or partial obstruction of the urinary tract.
  2. presence of active gastric/duodenal ulcer or gastrointestinal bleeding, of enteritis like Crohn's disease or ulcerative colitis, clinically confirmed coronary heart disease and/or cerebrovascular disease, cardiac insufficiency (NYHA II-IV), severe liver insufficiency, or severe renal insufficiency
  3. history of relevant CNS and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
  4. pathological ECG (12 standard leads)
  5. known allergic reactions to the active ingredient used, substituted benzimidazole or to other constituents of the pharmaceutical preparations
  6. subjects with severe allergies or multiple drug allergies
  7. positive results of the urine drug screen
  8. laboratory values out of normal range unless the deviation from normal is judged as not relevant for the study by the investigator
  9. positive anti-HIV-test, HBs-AG-test or anti-HCV-test
  10. lactose or fructose intolerance
  11. glucose-galactose malabsorption
  12. history of or current drug or alcohol dependence
  13. regular intake of alcoholic food or beverages of ≥ 40 g pure ethanol per day
  14. subjects who are on a diet which could affect the pharmacokinetics of the drug
  15. regular intake of caffeine containing food or beverages of ≥ 500 mg caffeine per day
  16. blood donation or other blood loss of more than 400 ml within the last two months prior to the start of the study
  17. participation in a clinical trial during the last two months prior to the start of the study
  18. subjects, who report a frequent occurrence of migraine attacks
  19. regular treatment with any systemically available medication (except hormonal replacement therapy e.g. L-thyroxine) within 14 days prior to the first administration of the study medication
  20. subjects suspected or known not to follow instructions

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Comparison of pharmacokinetic parameters of esomeprazole after single oral doses of Esomeprazole Mepha capsules (Test) and 40 mg Esomeprazole INexium MUPS tablets (Reference) under fasted and fed conditions. | April - June 2009

SECONDARY OUTCOMES:
Descriptive characterisation of safety and tolerability of the investigational products in the study population. | April - June 2009

CONTACTS AND LOCATIONS:
Overall Officials: Frank Donath, MD, Principal Investigator — SocraTec R&D GmbH
Locations (1):
- SocraTec R&D Probandenstation, Erfurt, Thuringia, Germany